CLINICAL TRIAL: NCT06054802
Title: The Influence of Perioperative Sleep Quality on Postoperative Pain Outcomes in Pediatric Patients Undergoing Knee Surgery
Brief Title: Perioperative Sleep Quality and Postoperative Pain Outcomes
Status: Enrolling by invitation | Type: Observational
Sponsor: Grant Heydinger (Other)
Responsible Party: Sponsor-Investigator, Grant Heydinger, Assistant Professor of Anesthesiology, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: STUDY00003629
Record Dates: First submitted 2023-09-20; First posted 2023-09-26 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Surgery; ACL Injury; Pain; Sleep
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ACL surgery: Pediatric subjects undergoing surgery for ACL repair.
  Interventions: Device: eCAP

INTERVENTIONS:
Device: eCAP — eCap™ has the look and feel of a regular prescription bottle and records real-time adherence data, tracking each opening with the date and time.

SUMMARY:
This is a prospective, observational cohort study that will examine how sleep quality impacts postoperative pain and opioid consumption for pediatric patients. The investigators will administer a questionnaire preoperatively to determine which patients have poor or good sleep quality. They will then compare postoperative pain and opioid use between groups for two weeks following surgery. For a secondary aim, investigators will use electronic medication vials (eCAP) to monitor participants' medication use at home and compare to self-reporting.

ELIGIBILITY:
Inclusion Criteria:

* able to read, understand, and speak English
* are undergoing ACL repair or reconstruction
* have availability of a mobile device/computer to receive text messages

Exclusion Criteria:

* < 10 or > 18 years of age
* have a history of sleep-disordered breathing including sleep apnea
* have a history of chronic pain or current opioid use
* have a history of developmental delay that would preclude study participation

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric/adolescent patients undergoing anterior cruciate ligament (ACL) repair or reconstruction at Nationwide Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | Baseline
  Pittsburgh Sleep Quality Index (PSQI) is a validated, self-report questionnaire that assesses sleep quality over a one-month period that takes five to ten minutes to complete. It offers seven component scores (e.g., subjective sleep quality, latency, duration, and efficiency) as well as a composite score that measures overall sleep quality. A total score greater than five yields a sensitivity of 89.6% and specificity of 86.5% (kappa = 0.75, p <0.001) in distinguishing good from poor sleepers.
Difference in opioid consumption between self-report and eCap | Days 1-14 post-op
  The eCAP Electronic Content Monitor (ECM) is a smart pill bottle used to monitor and improve medication adherence. When opened, an event is recorded, and the data is securely stored. The eCAP device timestamps medication usage and provides a visualization demonstrating how patients are taking medications, providing robust analytics. Subjects will also record each time they take an opioid pain medicine on a daily diary.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided